CLINICAL TRIAL: NCT00226161
Title: Chronic Pain After Inguinal Herniorrhaphy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 171178
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2005-09

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

INTERVENTIONS:
Procedure: Inguinal herniorrhaphy

SUMMARY:
The purpose of this study is to determine whether laparoscopic inguinal hernia repair leads to a lower incidence of chronic pain compared to open herniorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* Primary inguinal hernia

Exclusion Criteria:

* History of severe mental illness or chronic pain elsewhere

Ages: 18 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Dates: Start 2005-09; Primary Completion 2013-09; Study Completion 2013-09

PRIMARY OUTCOMES:
Chronic pain

SECONDARY OUTCOMES:
Recurrence of the hernia

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, professor,dr.med,chief consul, Study Director — Gentofte University Hospital
Locations (1):
- Department of Surgical Gastroenterology, Gentofte University Hospital,, Hellerup, Denmark